CLINICAL TRIAL: NCT00327314
Title: Non-Myeloablative Allogeneic Transplantation From Unrelated Donors in Multiple Myeloma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM 1641
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Last update posted 2006-12-28 (Estimated); Status verified 2006-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Transplantation; Stem Cell Transplantation

INTERVENTIONS:
Procedure: Transplantation
Procedure: Hematopoietic cell transplantation

SUMMARY:
The protocol aims at reducing transplant toxicity and mortality in patients with multiple myeloma.

DETAILED DESCRIPTION:
Primary end points are engraftment and non-relapse mortality. Secondary end points are disease response, overall survival, progression and event free survivals. Patient eligibility criteria.

Inclusion criteria included:

* Diagnosis of Durie-Salmon stage IIA-IIIB multiple myeloma
* Age > 18 and ≤ 65 years at the start of the donor search
* Presence of concurrent co-morbidities precluding myeloablative conditioning or refusal to undergo a conventional allogeneic transplant
* Capacity to give informed consent

Exclusion criteria included:

* Age > 65 years
* Karnofsky performance status score < 60%
* Progressive disease or stable disease for less than three months
* Central nervous system (CNS) involvement
* Left ventricular ejection fraction < 35% or symptomatic heart failure
* Poorly controlled hypertension
* Pulmonary dysfunction with diffusing capacity for carbon monoxide (DLCO) < 40% and/or need for continuous oxygen supplementation
* Abnormal liver disease with a serum bilirubin greater than twice normal or SGOT and/or SGPT greater than four times the upper limits of normal
* HIV positive patients
* Pregnancy
* Refusal to use contraceptive techniques during and for 12 months following treatment

Informed consent is obtained during study registration from each patient according to the Institutional Review Boards of the participating centers. The study is conducted according to the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Durie-Salmon stage IIA-IIIB multiple myeloma
* Age > 18 and ≤ 65 years at the start of the donor search
* Presence of concurrent co-morbidities precluding myeloablative conditioning or refusal to undergo a conventional allogeneic transplant
* Capacity to give informed consent

Exclusion Criteria:

* Age > 65 years
* Karnofsky performance status score < 60%
* Progressive disease or stable disease for less than three months
* Central nervous system involvement
* Left ventricular ejection fraction < 35% or symptomatic heart failure
* Poorly controlled hypertension
* Pulmonary dysfunction with diffusing capacity for carbon monoxide (DLCO) < 40% and/or need for continuous oxygen supplementation
* Abnormal liver disease with a serum bilirubin greater than twice normal or SGOT and/or SGPT greater than four times the upper limits of normal
* HIV positive patients
* Pregnancy
* Refusal to use contraceptive techniques during and for 12 months following treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-12; Study Completion 2006-10

CONTACTS AND LOCATIONS:
Overall Officials: Benedetto Bruno, MD, PhD, Principal Investigator — Divisione di Ematologia _ Azienda Ospedaliera S G Battista di Torino
Locations (1):
- Divisione Universitaria Ematologia Azienda Ospedaliera S G Battista, Torino, Italy